CLINICAL TRIAL: NCT05273476
Title: Augmentation of Keratinized Tissue Around Dental Implant With Combined Application of a Xenogeneic Collagen Matrix and the Free Gingival Graft : a Single Arm Clinical Trial
Brief Title: Augmentation of Keratinized Tissue Around Dental Implant With a Xenogeneic Collagen Matrix and the Free Gingival Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Dental Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Peihui Ding, Principal Investigator, The Dental Hospital of Zhejiang University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHZhejiangU-2022（023）
Record Dates: First submitted 2022-02-24; First posted 2022-03-10 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Inadequately Attached Gingiva

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- strip (Experimental): apically repositioned flap+ xenogeneic collagen matrix +free gingival graft
  Interventions: Procedure: apically repositioned flap+ xenogeneic collagen matrix +free gingival graft

INTERVENTIONS:
Procedure: apically repositioned flap+ xenogeneic collagen matrix +free gingival graft — Harvest a strip free gingival graft from the palate, then place it above apically repositioned flap and fix xenogeneic collagen matrix to the recipient bed

SUMMARY:
The purpose of this study is to compare the clinical effects of combined application of combined application of a xenogeneic collagen matrix and the free gingival graft in augmentation of keratinized tissue around dental implant by single arm clinical trial, compared with historical control group 1:application of a xenogeneic collagen matrix,and historical control group 2:application of the free gingival graft.

DETAILED DESCRIPTION:
The purpose of this study is to compare the clinical effects of combined application of a xenogeneic collagen matrix and the free gingival graft in augmentation of keratinized tissue around dental implant by single arm clinical trial, compared with historical control group 1:application of a xenogeneic collagen matrix,and historical control group 2:application of the free gingival graft. This study designed a single arm clinical trial. The included patients will all be treated with apical repositioned flap with a xenogeneic collagen matrix and the free gingival graft. The width of keratinized mucosa, thickness of keratinized mucosa, gingival index, probing depth will be measured before surgery and at 2, 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Aged >=18 years and periodontally and systemically healthy;
2. Presence of at least one site with <=2 mm of keratinized tissue; associated with a shallow vestibule in the edentulous region after implant surgery (no more than three consecutive implants);
3. Need of keratinized tissue augmentation for aesthetic purpose and/or functional reasons;
4. Full mouth probing depths <=5mm;
5. Full-mouth plaque score (FMPS) and full-mouth bleeding score (FMBS) <=15%;
6. Be able to comply with all procedures related to the study.

Exclusion Criteria:

1. Smoking;
2. Pregnant or lactating women;
3. Untreated periodontal disease;
4. Presence of systemic disorders (diabetes, heart disease, tumor or any other condition that could contraindicate periodontal surgery);
5. Use of medications (immunosuppressants, phenytoin, or anything else that might affect mucosal healing and repair);
6. Under radiotherapy;
7. Allergy to the collagen;
8. Previous mucogingival surgery in the area.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
change from baseline keratinized mucosa width at 2 and 6 months | baseline, at 2,6 months
  measured from the mucogingival junction to the mucosa margin or the zenith of alveolar ridge at the mid-buccal aspect of each implant using a periodontal probe (UNC15)

SECONDARY OUTCOMES:
change from baseline keratinized mucosa thickness at 2 and 6 months | baseline, at 2,6 months
  measured at the middle point of an apical-coronal direction at the mid-buccal aspect using an endodontic file with a rubber stop
change from baseline Gingival index at 2 and 6 months | baseline, at 2,6 months
  assessed at four gingival sites of each implant (mesio-labial/buccal, mid-labial/buccal, disto-labial/buccal, and palatal/lingual) . Indicated by numbers, 0: normal gingiva; 1: slightly edematous gingiva that does not bleed on probing; 2: edematous gingiva that bleeds on probing; 3: gingiva that has a tendency to bleed spontaneously or ulcerate.
change from baseline probing depth at 2 and 6 months | baseline, at 2,6 months
  measured at six sites of each implant (mesio-labial/buccal, mid-labial/buccal, disto-labial/buccal, mesio-palatal/lingual, mid-palatal/lingual, and disto-palatal/lingual) using a periodontal probe (UNC15)
Post-operative pain | at 1 week after surgery
  evaluated using a visual analog scale (VAS) ranging from 0 to 10 (0 = no pain and 10 = worst pain imaginable)
change from 2 months patient satisfaction at 6 months | at 2 and 6 months post operation
  using a visual analog scale (VAS) ranging from 0 to 10 (0 = extremely dissatisfied and 10 = extremely satisfied)
dosage of postoperative analgesic drugs | at 1 week after surgery
  dosage of postoperative analgesic drugs that patients take after surgery
operation time | during the surgery
  measured from the start of the first incision to the end of the last suture
esthetic score | at 6 months post operation
  assessed by judging on the colour, contour, and texture of the surgical sites
change from baseline depth of recession at 2 and 6 months | baseline, at 2,6 months
  The distance from the implant margin to the gingival margin was measured with a periodontal probe
change from baseline width of recession at 2 and 6 months | baseline, at 2,6 months
  The proximal and distal level of soft tissue retraction at the top of implant was measured by periodontal probe

CONTACTS AND LOCATIONS:
Overall Officials: Peihui Ding, Doctor, Principal Investigator — The Affiliated Stomatology Hospital of Zhejiang University School of Medicine
Locations (1):
- The Affiliated Stomatology Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No